CLINICAL TRIAL: NCT02814526
Title: Therapeutic Effects of Exercise in Adults With Amnestic Mild Cognitive Impairment (MCI)
Brief Title: Exercise in Adults With Mild Memory Problems
Acronym: EXERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADC-041-EX; U19AG010483-22 (NIH)
Record Dates: First submitted 2016-06-02; First posted 2016-06-27 (Estimated); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment; Cognitive Decline; Memory Impairment
Keywords: exercise
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic (Experimental): Moderate/high intensity aerobic exercise will involve training at 70-80% heart rate reserve for 30 min, with an additional 10 minutes for warm-up and 5 minutes for cool-down, 4 times per week, for 12 months while supervised twice per week by a study-certified trainer at a participating YMCA .
  Interventions: Behavioral: Aerobic exercise
- Stretching/balance/range of motion (Active Comparator): The stretching/balance/range of motion program will involve exercise at or below 35% heart rate reserve for 30 min, with an additional 10 minutes for warm up and 5 minutes for cool-down, 4 times per week, for 12 months while supervised twice per week by a study-certified trainer at a participating YMCA.
  Interventions: Behavioral: Stretching/balance/range of motion exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Moderate/high intensity aerobic exercise will involve training at 70-80% heart rate reserve for 30 min, with an additional 10 minutes for warm-up and 5 minutes for cool-down, 4 times per week, for 12 months while supervised twice per week by a study-certified trainer at a participating YMCA .
  Arms: Aerobic
Behavioral: Stretching/balance/range of motion exercise — The stretching/balance/range of motion program will involve exercise at or below 35% heart rate reserve for 30 min, with an additional 10 minutes for warm up and 5 minutes for cool-down, 4 times per week, for 12 months while supervised twice per week by a study-certified trainer at a participating YMCA.
  Arms: Stretching/balance/range of motion

SUMMARY:
This study evaluates the effects of physical exercise on cognition, functional status, brain atrophy and blood flow, and cerebrospinal fluid biomarkers of Alzheimer's disease in adults with a mild memory impairment.

Half of participants will participate in a stretching-balance-range of motion exercise program, while the other half will participate in a moderate/high aerobic training program.

DETAILED DESCRIPTION:
Overall Study Design:

The EXERT trial was a multicenter phase 3 randomized, single-blind study that examined the effects of aerobic exercise on cognition, functional status, whole and regional cerebral blood flow, and cerebrospinal fluid biomarkers of Alzheimer's disease in approximately 300 adults with amnestic MCI. EXERT included an 18-month behavioral intervention trial, with a 12-month supervised exercise intervention phase with its primary endpoints, followed by a 6-month unsupervised exercised phase.

Subject Populations and Group Assignments:

The study population included male and female subjects aged 65 to 89 diagnosed with test scores and clinical ratings consistent with amnestic Mild Cognitive Impairment (MCI).

Assignment to study groups:

involved randomization to either treatment or active control, and study staff performing assessments were blinded to intervention assignment to maintain the single-blind structure of the trial.

Participants were to complete EXERT interventions at participating YMCAs located near the selected clinic sites across the U.S. The YMCA provided 18-month memberships at no cost to participants. In the first 12 months, a study-certified YMCA Trainer supervised all participants for the first 8 exercise sessions completed (weeks 1 and 2), and for 2 of 4 weekly sessions thereafter through Month 12. At Month 12, participants transitioned to independent exercise and were instructed to continue their assigned exercise programs for the final 6 months of the study without supervision. To encourage adherence and optimize cost efficiency, Trainers provided supervision to small groups of participants (2-4 individuals) randomized to the same intervention whenever possible. Compliance was evaluated using multiple mechanisms including heart rate monitoring, participant ratings of perceived exertion, entries in participants' Physical Activity Logs, Trainer assessment of effort, and weekly data review by the YMCA-Project Manager (Y-PM) and the Intervention Oversight Team (includes the Project Directors, Wake Forest team of exercise trial specialists, and Y-USA). These mechanisms provided multiple and regular opportunities to discuss participant progress, identify and resolve barriers, and encourage high levels of adherence to study protocols. The Intervention Oversight Team had the necessary expertise to successfully accomplish this objective in EXERT.

ELIGIBILITY:
Inclusion Criteria

1. Age between 65 and 89 years old, inclusive
2. MMSE: ≥24 for participants with 13 or more years of education; ≥22 for participants with 12 or fewer years of education
3. Global CDR score of 0.5 with a memory score of at least 0.5
4. Profile of test scores and clinical ratings is consistent with amnestic mild cognitive impairment
5. Speaks English fluently
6. Visual and auditory acuity adequate for cognitive testing
7. Completed at least 6 years of formal education or work history sufficient to exclude mental retardation
8. Has an informant who knows the participant well, has regular contact, and is available to accompany the participant to clinic visits or complete study partner assessments remotely.
9. Sedentary or underactive, determined by responses to the staff-administered EXERT Telephone Assessment of Physical Activity (TAPA) survey
10. Willing to be randomized to either intervention group and to complete the assigned activities as specified for 18 months
11. Willing and able to reliably travel to the identified YMCA, 4 times per week for 18 months
12. Ability to safely participate in either intervention and complete the 400 m Walk Test within 15 min without sitting or use of any assistance
13. Plans to reside in the area for at least 18 months
14. For planned travel, total time away must be no more than 2 months over the course of the study, and no more than 1 month at any one time; participants must be willing to continue the assigned exercise program if travelling out of the area for more than 1 week
15. In overall good general health with no disease or planned surgery that could interfere with study participation
16. Modified Hachinski ≤4
17. Stable use of cholinesterase inhibitors, memantine, vitamin E, estrogens, aspirin (81 300 mg daily), beta-blockers, or cholesterol-lowering agents for 12 weeks prior to screening (important for biomarker analyses)
18. Stable use of antidepressants lacking significant anticholinergic side effects for 4 weeks prior to screening as long as the participant does not meet DSM V criteria for major depression currently or in the last 12 months; GDS scores are to be used to inform clinical decisions but there is no specified cut-off score for inclusion
19. When applicable, willing to complete 4-week washout of psychoactive medications, including disallowed antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, and willing to avoid these medications for the duration of the trial
20. Able to complete all baseline assessments

Exclusion Criteria

1. Any significant neurologic disease, other than MCI, including any form of dementia, Parkinsons disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma with persistent neurologic sequelae or known structural brain abnormalities
2. Sensory or musculoskeletal impairment sufficient to preclude successful and safe completion of the intervention or assessment protocols; must be able to walk safely and unassisted on a treadmill
3. Contraindications for MRI studies, including claustrophobia, metal (ferromagnetic) implants, or cardiac pacemaker
4. Brain MRI at screening shows evidence of infection, infarction, or other clinically significant focal lesions, including multiple lacunes in prefrontal or critical memory regions; inconclusive findings may be subject to review by the ADCS Imaging Core
5. History of major depression or bipolar disorder (DSM V criteria), psychotic features, agitation or behavioral problems within the last 12 months
6. History of schizophrenia, as per DSM V criteria
7. History of alcohol or substance abuse or dependence within the past 2 years, as per DSM V criteria
8. Currently consumes more than 3 alcoholic drinks per day
9. Clinically significant or unstable medical condition, including uncontrolled hypertension or significant cardiac, pulmonary, hematologic, renal, hepatic, gastrointestinal, endocrine, metabolic or other systemic disease in the opinion of clinic medical personnel that may put the participant at increased risk, influence the results or compromise the participants ability to participate in the study (treated atrial fibrillation for more than 1 year or occasional premature ventricular contractions on ECG are not exclusions)
10. History in the last 6 months of myocardial infarction, coronary artery angioplasty, bypass grafting, or STENT placement
11. History in the last 3 months of transient ischemic attack or small vessel stroke (if more than 3 months, small vessel stroke with no residual effects are permitted)
12. Expected joint replacement surgery within the next 18 months
13. History within the last 5 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen posttreatment
14. Hemoglobin A1c >7.0
15. Clinically significant abnormalities in screening laboratory blood tests: low B12 is exclusionary, unless follow-up labs (homocysteine [HCY] and methylmalonic acid [MMA]) indicate that it is not physiologically significant
16. Current or past use of insulin to treat type 2 diabetes (other diabetes medications are acceptable if hemoglobin A1c ≤7)
17. Current use (within 60 days of screening) of psychoactive medications including tricyclic antidepressants, antipsychotics, mood-stabilizing psychotropic agents (e.g. lithium salts), psychostimulants, opiate analgesics, antiparkinsonian medications, anticonvulsant medications (except gabapentin and pregabalin for non-seizure indications), systemic corticosteroids, or medications with significant central anticholinergic activity. Limited use of antipsychotics (quetiapine ≤ 50mg/day or risperidone ≤ 0.5mg/day), and non-chronic use of opiate analgesics on an as needed basis is permitted; such medications must be avoided for 8 hours before clinic assessments
18. Chronic use of anxiolytics or sedative hypnotics except as follows: use of benzodiazepines for treatment on an as-needed basis for insomnia or daily dosing of anxiolytics is permitted; medications must be avoided for 8 hours before clinic assessments
19. Previous or current treatment involving active immunization against amyloid
20. Previous treatment with approved or investigational agents with anti-amyloid properties or passive immunization against amyloid are prohibited 12 months prior to screening and for the duration of the trial; treatment with other investigational agents are prohibited 3 months prior to screening and for the duration of the trial
21. For LP, current use of anticoagulants such as Coumadin, Plavix, or high dose Vitamin E
22. For LP, current blood clotting or bleeding disorder, or significantly abnormal prothrombin time (PT) or partial thromboplastin time (PTT) at screening
23. For LP, presence of physical distortions due to spinal surgery, severe degenerative joint disease or deformity, or obesity that could interfere with CSF collection (as per investigator judgment)
24. Participants whom the PI deems otherwise ineligible

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 296 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Feldman, MDCM FRCP(C), Principal Investigator — Alzheimer's Disease Cooperative Study (ADCS)
Locations (14):
- United States (14):
  - University of California, Irvine, Irvine, California
  - VAPAHCS / Stanford University School of Medicine, Palo Alto, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Great Lakes Clinical Trials (Andersonville), Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of North Texas Health Science Center, Fort Worth, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is integral to the ADCS's mission to develop and execute innovative clinical trials focused on interventions that may prevent, delay, or treat the expression of Alzheimer's disease and related dementias. The ADCS is committed to sharing resources and tools, including data, biospecimens, trial designs, outcome and analysis measures following NIH guidelines.
  DATA SHARING: The ADCS Data and Sample Sharing Committee (DSSC) grants access to de-identified data to individuals who complete the request process and agree to the conditions in an ADCS/UCSD Data Use Agreement (DUA). After approval and receipt of the fully executed DUA, applicants are authorized to acquire data. Non-compliance with the DUA, including the requirement to provide requested updates will jeopardize further access to data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01 March 2023
Access Criteria: Data requestors must complete an ADCS data and sample sharing request form. Upon approval, requestors must complete a data use agreement prior to accessing the data.
URL: https://www.adcs.org/data-sharing/

REFERENCES:
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Plymate SR, Fishel MA, Watson GS, Cholerton BA, Duncan GE, Mehta PD, Craft S. Effects of aerobic exercise on mild cognitive impairment: a controlled trial. Arch Neurol. 2010 Jan;67(1):71-9. doi: 10.1001/archneurol.2009.307. PMID 20065132
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Colcombe SJ, Erickson KI, Scalf PE, Kim JS, Prakash R, McAuley E, Elavsky S, Marquez DX, Hu L, Kramer AF. Aerobic exercise training increases brain volume in aging humans. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1166-70. doi: 10.1093/gerona/61.11.1166. PMID 17167157
- [Background] Voss MW, Prakash RS, Erickson KI, Basak C, Chaddock L, Kim JS, Alves H, Heo S, Szabo AN, White SM, Wojcicki TR, Mailey EL, Gothe N, Olson EA, McAuley E, Kramer AF. Plasticity of brain networks in a randomized intervention trial of exercise training in older adults. Front Aging Neurosci. 2010 Aug 26;2:32. doi: 10.3389/fnagi.2010.00032. eCollection 2010. PMID 20890449
- [Background] Colcombe SJ, Erickson KI, Raz N, Webb AG, Cohen NJ, McAuley E, Kramer AF. Aerobic fitness reduces brain tissue loss in aging humans. J Gerontol A Biol Sci Med Sci. 2003 Feb;58(2):176-80. doi: 10.1093/gerona/58.2.m176. PMID 12586857
- [Background] Burns JM, Cronk BB, Anderson HS, Donnelly JE, Thomas GP, Harsha A, Brooks WM, Swerdlow RH. Cardiorespiratory fitness and brain atrophy in early Alzheimer disease. Neurology. 2008 Jul 15;71(3):210-6. doi: 10.1212/01.wnl.0000317094.86209.cb. PMID 18625967
- [Result] Nichol KE, Poon WW, Parachikova AI, Cribbs DH, Glabe CG, Cotman CW. Exercise alters the immune profile in Tg2576 Alzheimer mice toward a response coincident with improved cognitive performance and decreased amyloid. J Neuroinflammation. 2008 Apr 9;5:13. doi: 10.1186/1742-2094-5-13. PMID 18400101
- [Derived] Shadyab AH, Aslanyan V, Jacobs DM, Salmon DP, Morrison R, Katula JA, Jin S, Thomas RG, LaCroix AZ, Pa J, Cotman CW, Feldman HH, Baker LD; ADCS EXERT Study Group. Effects of exercise versus usual care on older adults with amnestic mild cognitive impairment: EXERT versus ADNI. Alzheimers Dement. 2025 Apr;21(4):e70118. doi: 10.1002/alz.70118. PMID 40271887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Academic Institutions and participating Y-USA Centers across the nation. Recruitment for the overall study began June 2016 and ended in October 2021. This study consisted of a four week screening period, followed by 12 months of supervised exercise (the ITT period), and an additional 6 month unsupervised exercise period.
Pre-assignment Details: Screening duration: From signed consent up to 4 weeks. At baseline visit, participants are randomized to trial arms. A total of 532 participants consented to participate in the trial. Of these consented, 236 participants were screening failures. 296 participants were assigned/randomized to the trial.
Period: Overall Study
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Started | 148 | 148
Completed (Completed = number of participants randomized to AX or SBR and completed 12 months of supervised exercise sessions) | 115 | 118
Not Completed | 33 | 30
Not completed — Adverse Event | 4 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 4
Not completed — non site physician decision | 1 | 0
Not completed — participant noncompliance | 1 | 1
Not completed — Withdrawal by Subject | 20 | 14
Not completed — safety risk | 2 | 1
Not completed — early termination-study terminated | 1 | 2
Not completed — Other | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic | Stretching/Balance/Range of Motion | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.26 (5.71) | 74.65 (6.23) | 74.46 (5.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 84 | 169
  Male | 63 | 64 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 142 | 145 | 287
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 127 | 129 | 256
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 148 | 148 | 296
Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination is a brief mental status exam and widely used dementia screening instrument. It evaluates orientation to time and place, memory, attention, language, and visuospatial ability. Range: 0-30; a lower score indicates greater impairment.
  units on a scale | 27.92 (1.91) | 28.03 (1.83) | 27.97 (1.87)
Alzheimer's Disease Assessment Scale - Cognitive Subscale 13 (ADAS-Cog 13) [Mean (Standard Deviation); unit: units on a scale] — ADAS-Cog13 is a structured scale that evaluates memory (immediate and delayed word recall; immediate word recognition), receptive and expressive language, orientation, ideational praxis (preparing a letter for mailing), constructional praxis (copying figures), and attention (number cancellation). Ratings of spoken language, language comprehension, word finding difficulty, and ability to remember test instructions also are obtained. Range: 0-85; higher scores indicate greater impairment. Population: Baseline scores for this measure only available for 294 participants out of 296 total baselined.
  units on a scale
    number analyzed (Participants) | 147 | 147 | 294
    (all) | 13.82 (6.62) | 14.23 (6.81) | 14.02 (6.71)
Clinical Dementia Rating - Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: units on a scale] — CDR-SB is a composite rating of cognition and everyday function which incorporates both informant input and direct assessment of performance. It assesses through semi-structured interview three cognitive domains (memory, orientation, and judgement/problem solving) and three everyday functional domains (community affairs, home and hobbies, personal care). Level of impairment in each of the six domains is rated from none (score=0) to severe (score=3). The six domain scores are then summed to create the CDR-SB. Range 0-18; higher scores indicate greater impairment. Population: Baseline scores for this measure only available for 295 participants out of 296 total baselined.
  units on a scale
    number analyzed (Participants) | 148 | 147 | 295
    (all) | 1.43 (0.84) | 1.57 (0.87) | 1.5 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: ADAS-Cog-Exec Global Composite
Description: The ADAS-Cog-Exec Composite is a weighted sum of standardized (Z-score) change on subtests from the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog13; Immediate and Delayed Word Recall, Orientation, and Number Cancellation); box scores for the cognitive components of the Clinical Dementia Rating Scale (Memory, Orientation, Judgement & Problem Solving); and additional tests requiring executive function (Trail Making Test A & B, Digit Symbol Substitution, Category Fluency). See https://doi.org/10.1002/trc2.12059 for a detailed description regarding the development and validation of the ADAS-Cog-Exec.
  Change for the analysis of this primary outcome was calculated comparing the average of scores from month 6 and month 12 to baseline. The theoretical range for the ADAS-Cog-Exec is -3.00 to +3.00 in EXERT, with higher scores indicating improvement in cognitive function from baseline.
Time Frame: Baseline to mean (Mo 6, Mo 12)
Population: Modified Intent-to-Treat (mITT) Population: Includes all eligible participants who (1) began the exercise intervention (Intervention Session 1) and (2) completed at least one post-baseline assessment for the primary analysis at Month 6 or Month 12.
  All consented randomized participants are grouped according to the treatment assigned at randomization, regardless of any protocol violations.
Measure: Least Squares Mean (Standard Error); unit: Change score
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 124 | 126
Change score | -0.146 (0.063) | -0.068 (0.063)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.29, Regression, Linear; Mean Difference (Net) = 0.078

2. Secondary Outcome: ADAS-Cog-Exec Global Composite in Subset Population
Description: as for outcome 1
Time Frame: Baseline to mean (Mo 6, Mo 12)
Population: Subset of participants who had the opportunity to complete a full 12 months of the study (i.e., 12 months of exercise and the 12 Month outcome assessments) before the COVID-19 pandemic affected trial conduct.
Measure: Least Squares Mean (Standard Error); unit: Change score
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 70 | 73
Change score | -0.18 (0.080) | -0.15 (0.076)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.74, Regression, Linear; Mean Difference (Net) = 0.031

3. Secondary Outcome: Executive Function Composite Score
Description: The Executive Function Composite is the average standardized (Z-score) change on eight measures requiring attention and executive control: Trail Making, Part B; Digit Symbol Substitution; Category Fluency; Letter Fluency; Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog13) Number Cancellation; NIH Toolbox Flanker; NIH Toolbox Dimension Change Card Sort, and Cogstate One Back.
  Change for analysis of this secondary outcome was calculated comparing the average of scores from month 6 and month 12 to baseline. The theoretical range for the Executive Function Composite is -3.00 to +3.00, with higher scores indicating improvement in executive function from baseline.
Time Frame: Baseline to mean (Mo 6, Mo 12)
Measure: Least Squares Mean (Standard Error); unit: Change in score
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 109 | 112
Change in score | -0.02903 (0.03303) | -0.03847 (0.03246)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.8284, Regression, Linear; Mean Difference (Net) = -0.009447

4. Secondary Outcome: Episodic Memory Composite Score
Description: The Episodic Memory Composite is the average standardized (Z-score) change on five measures of memory: Immediate and Delayed Word Recall from the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog13); Cogstate Face-Name Associative Memory; Cogstate Behavioral Pattern Separation of Objects; and Cogstate One Card Learning.
  Change for analysis of this secondary outcome was calculated comparing the average of scores from month 6 and month 12 to baseline. The theoretical range for the Episodic Memory Composite is -3.00 to +3.00, with higher scores indicating improvement in episodic memory from baseline.
Time Frame: Baseline to mean (Mo 6, Mo 12)
Measure: Least Squares Mean (Standard Error); unit: Change in score
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 97 | 104
Change in score | 0.005859 (0.04137) | -0.014384 (0.03997)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.7086, Regression, Linear; Mean Difference (Net) = -0.02024

5. Secondary Outcome: Volumetric Magnetic Resonance Imaging (MRI) of Hippocampus
Description: Assessment of volumetric change in the hippocampus region of the brain, measured by structural Magnetic Resonance Imaging (MRI), comparing MRI scans taken at baseline and month 12. Scans are compared and analyzed to give a percent deformation between timepoints.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percent deformation
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 90 | 93
percent deformation | -0.66 (1.12) | -0.343 (0.98)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.06, Regression, Linear; Mean Difference (Net) = 0.29

6. Secondary Outcome: Volumetric Magnetic Resonance Imaging (MRI) of Prefrontal Composite Region
Description: Assessment of volumetric change in prefrontal composite regions of the brain, measured by structural Magnetic Resonance Imaging (MRI), comparing MRI scans taken at baseline and month 12. The prefrontal composite includes: superior frontal, caudal-middle frontal, rostral-middle frontal, pars opercularis, and pars triangularis regions. Scans are compared and analyzed to give a percent deformation between timepoints.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percent deformation
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 90 | 93
percent deformation | -0.34 (1.36) | -0.51 (1.11)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.33, Regression, Linear; Mean Difference (Net) = -0.17

7. Secondary Outcome: Volumetric Magnetic Resonance Imaging (MRI) of AD Signature Composite Region
Description: Assessment of volumetric change in Alzheimer's Disease (AD) signature regions of the brain, measured by structural Magnetic Resonance Imaging (MRI), comparing MRI scans taken at baseline and month 12. The AD signature composite includes: parahippocampus, fusiform, inferior temporal, middle temporal, and inferior-parietal regions. Scans are compared and analyzed to give a percent deformation between timepoints.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percent deformation
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 90 | 93
percent deformation | -0.612 (1.02) | -0.643 (0.951)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.49, Regression, Linear; Mean Difference (Net) = -0.10

8. Secondary Outcome: Arterial Spin Labeling (ASL) Magnetic Resonance Imaging (MRI) of Hippocampus
Description: Assessment of change in blood flow activity in the hippocampus region of the brain, measured using Arterial Spin Labeling (ASL) magnetic resonance imaging (MRI) scans. Scans taken at baseline and month 12 are compared and analyzed to assess change in blood flow between the timepoints. The unit of cerebral blood flow from ASL is ml/100g/min, which means the amount of blood flow into 100g of tissue during one minute.
Time Frame: Baseline to 12 Months
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 73 | 66
ml/100g/min | 0.07 (0.42) | 0.01 (0.224)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.61, Regression, Linear; Mean Difference (Net) = -0.02

9. Secondary Outcome: Arterial Spin Labeling (ASL) Magnetic Resonance Imaging (MRI) of Prefrontal Composite Region
Description: Assessment of change in blood flow activity in the prefrontal composite regions of the brain, measured using Arterial Spin Labeling (ASL) magnetic resonance imaging (MRI) scans. The prefrontal composite includes: superior frontal, caudal-middle frontal, rostral-middle frontal, pars opercularis, and pars triangularis regions. Scans taken at baseline and month 12 are compared and analyzed to assess change in blood flow. The unit of cerebral blood flow from ASL is ml/100g/min, which means the amount of blood flow into 100g of tissue during one minute.
Time Frame: Baseline to 12 Months
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 73 | 66
ml/100g/min | 0.04 (0.31) | 0.03 (0.29)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.78, Regression, Linear; Mean Difference (Net) = -0.01

10. Secondary Outcome: Arterial Spin Labeling (ASL) Magnetic Resonance Imaging (MRI) of AD Signature Composite Region
Description: Assessment of change in blood flow activity in the Alzheimer's Disease (AD) signature regions of the brain, measured using Arterial Spin Labeling (ASL) magnetic resonance imaging (MRI) scans. The AD signature composite includes: parahippocampus, fusiform, inferior temporal, middle temporal, and inferior-parietal regions. Scans taken at baseline and month 12 are compared and analyzed to assess change in blood flow. The unit of cerebral blood flow from ASL is ml/100g/min, which means the amount of blood flow into 100g of tissue during one minute.
Time Frame: Baseline to 12 Months
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 73 | 66
ml/100g/min | 0.05 (0.23) | 0 (0.25)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.31, Regression, Linear; Mean Difference (Net) = -0.04

11. Secondary Outcome: Ratio of AD Biomarkers in Blood
Description: Change in ratio of plasma amyloid beta peptides in blood plasma from baseline to12 months. A lower ab42/ab40 ratio in plasma is associated with a higher risk of dementia.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Change in ratio
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 103 | 111
Change in ratio | 0.00001 (0.0185) | -0.00062 (0.01119)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.817, Regression, Linear; Mean Difference (Net) = -0.0005

12. Secondary Outcome: AD Biomarkers in CSF (ab42/ab40)
Description: Change in ratio of amyloid beta peptides in cerebrospinal fluid (CSF) from baseline to 12 months. A lower ab42/ab40 ratio is associated with a higher risk of dementia.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Change in ratio
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 14 | 10
Change in ratio | -0.00348 (0.00784) | -0.00413 (0.00611)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.64, Regression, Linear; Mean Difference (Net) = 0.0020

13. Secondary Outcome: AD Biomarkers in CSF (ab42/Tau)
Description: Change in ratio of key peptides in cerebrospinal fluid (CSF) from baseline to 12 months. A lower ab42/tau ratio is associated with a higher risk of dementia.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Change in ratio
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 14 | 10
Change in ratio | -0.22 (0.445) | -0.299 (0.729)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.97, Regression, Linear; Mean Difference (Net) = -0.01

14. Secondary Outcome: AD Biomarkers in CSF (ab42/P-tau)
Description: Change in ratio of key peptides in cerebrospinal fluid (CSF) from baseline to 12 months. A lower ab42/p-tau ratio is associated with a higher risk of dementia.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Change in ratio
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
Number analyzed (Participants) | 14 | 10
Change in ratio | -2.48 (2.70) | -3.39 (5.47)
Statistical Analysis 1: Comparison: Aerobic vs Stretching/Balance/Range of Motion; Test type: Superiority; p = 0.94, Regression, Linear; Mean Difference (Net) = -0.17

15. Other Pre Specified Outcome: Intervention Effects on Secondary Outcomes in a Subset of Participants Who Completed 12 Months of the Study Prior to the COVID-19 Pandemic.
Description: To examine intervention effects on secondary outcomes listed above in participants who had the opportunity to complete a full 12 months of the study before the pandemic affected trial conduct.
Time Frame: 12 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploratory Magnetic Resonance Imaging (MRI) Volumes and Perfusion and Individual AD Biomarkers in CSF and Blood Measures
Description: To test whether 12 months of aerobic exercise, relative to the control, favorably affects MRI whole brain, ventricular and entorhinal volumes; perfusion in whole brain, gray matter and white matter; and individual AD biomarkers in CSF (ab42, ab40, total tau, p-tau, BDNF) and blood (ab42, ab40).
Time Frame: 12 Months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Clinical Dementia Rating Scale-Sum of Boxes (CDR) and Alzheimers Disease Assessment Scale-Cognitive 13-item (ADAS-Cog13)
Description: To test whether 12 months of aerobic exercise, relative to the control, reduces clinical ratings of cognitive impairment as measured by the CDR Sum of Boxes, and total score on the ADAS Cog13.
Time Frame: 12 Months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Measures of Cognitive Function and Well-being Including (1) ADCS-ADL-MCI); (2) BRIEF-A; (3) GDS; (4) NPI; SF-36; EuroQol: 5-Item Health Questionnaire; (5) CCI: Cognitive Change Index); and (6) Study Partner Self-Assessment
Description: To test whether 12 months of aerobic exercise, relative to the control, improves self-report measures of cognitive function and well-being, including (1) daily living skills (ADCS-Activities of Daily Living-MCI); (2) BRIEF-A: Behavior Rating Inventory of Executive Function-Adult Version); (3) mood (GDS); (4) health-related quality of life (NPI: Neuropsychiatric Inventory; SF-36: 36-Item Short Form Health Survey; EuroQol: 5-Item Health Questionnaire); (5) subjective memory concerns (CCI: Cognitive Change Index); and (6) Study Partner Self-Assessment Questionnaire
Time Frame: 12 Months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: ADAS-Cog-Exec, Executive Function, and Episodic Memory Composites
Description: To examine enduring cognitive effects (measured by ADAS-Cog-Exec, Executive Function and Episodic Memory Composites) of the intervention following a 6-month extension (through Month 18) when the prescribed exercise is continued without supervision.
Time Frame: 18 Months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Subgroup Treatment Responder Analyses
Description: To explore whether sex, age, baseline AD biomarker profile in CSF (ab42/ab40, ab42/tau, ab42/p-tau) and blood (ab42/ab40), and ApoE4 genotype (e4+, e4-) predict treatment response.
Time Frame: 12 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data is collected from the time of consent through the 12 month supervised exercise period and through the following 6 month unsupervised exercise period.
Description: Adverse Event (AE)reporting begins at the time of consent. Collection of AEs was done through participant reporting using both systematic and non-systematic assessment of AEs.
  Systematic collection of AEs occurred at each scheduled participant visit capturing the events in source documents and electronic case report forms (eCRF).
  Non-systematic AE reporting, spontaneous reporting by participant between visits, was also implemented.
Arm/Group | Aerobic | Stretching/Balance/Range of Motion
All-Cause Mortality (participants affected / at risk) | 1/148 | 2/148
Serious Adverse Events (participants affected / at risk) | 23/148 | 23/148
Other Adverse Events (participants affected / at risk) | 148/148 | 148/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic (N=148) | Stretching/Balance/Range of Motion (N=148)
Cardiac disorders (Cardiac disorders) | 4 | 3
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1
Infections and infestations (Infections and infestations) | 5 | 4
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 | 2
Investigations (Investigations) | 0 | 2
Neoplasms benign, malignant and unspecified (cysts and polyps) 1 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nervous system disorders (Nervous system disorders) | 2 | 4
Psychiatric disorders (Psychiatric disorders) | 2 | 0
Renal and urinary disorders (Renal and urinary disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders 0 1 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Surgical and medical procedures 4 4 (Surgical and medical procedures) | 4 | 4
Vascular disorders 1 0 (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic (N=148) | Stretching/Balance/Range of Motion (N=148)
Cardiac disorders 11 9 (Cardiac disorders) | 11 | 9
Ear and labyrinth disorders (Ear and labyrinth disorders) | 4 | 1
Endocrine disorders (Endocrine disorders) | 1 | 0
Eye disorders (Eye disorders) | 4 | 4
Gastrointestinal disorders (Gastrointestinal disorders) | 9 | 19
General disorders and administration site conditions (General disorders) | 13 | 15
Immune system disorders (Immune system disorders) | 3 | 3
Infections and infestations (Infections and infestations) | 60 | 51
Injury, poisoning and procedural complications 76 59 (Injury, poisoning and procedural complications) | 76 | 59
Investigations 6 8 (Investigations) | 6 | 8
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 | 0
Musculoskeletal and connective tissue disorders 78 70 (Musculoskeletal and connective tissue disorders) | 78 | 70
Neoplasms benign, malignant and unspecified (cysts and polyps) 6 6 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Nervous system disorders 18 29 (Nervous system disorders) | 18 | 29
Psychiatric disorders 4 6 (Psychiatric disorders) | 4 | 6
Renal and urinary disorders 4 6 (Renal and urinary disorders) | 4 | 6
Reproductive system and breast disorders 1 0 (Reproductive system and breast disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders 8 3 (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Skin and subcutaneous tissue disorders 8 2 (Skin and subcutaneous tissue disorders) | 8 | 2
Surgical and medical procedures 19 17 (Surgical and medical procedures) | 19 | 17
Vascular disorders 9 3 (Vascular disorders) | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT02814526/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT02814526/SAP_001.pdf
  • Informed Consent Form (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT02814526/ICF_002.pdf